CLINICAL TRIAL: NCT04783649
Title: Clinical Validation of Cervical Cancer Screening Methods in St. Petersburg, Russia
Brief Title: Clinical Validation of Cervical Cancer Screening Methods
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: N.N. Petrov National Medical Research Center of Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: CC-001
Record Dates: First submitted 2021-03-02; First posted 2021-03-05 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: Cervical Cancer; Cervical Dysplasia; Human Papilloma Virus
MeSH Terms: conditions — Uterine Cervical Neoplasms; Uterine Cervical Dysplasia | interventions — Colposcopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Cytology and biopsy samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- High risk group: Women in the age group between 25 and 65 years old without prior history of malignancy referred to colposcopy
  Interventions: Diagnostic Test: Papanicolaou cytological test; Diagnostic Test: Local cytological test (H&E stain); Diagnostic Test: Validated HPV DNA Test; Diagnostic Test: Local HPV test; Diagnostic Test: Colposcopy
- Population sample: A population sample of women in the age group between 25 and 65 years old from several primary healthcare facilities to primary cervical screening
  Interventions: Diagnostic Test: Papanicolaou cytological test; Diagnostic Test: Local cytological test (H&E stain); Diagnostic Test: Validated HPV DNA Test; Diagnostic Test: Local HPV test

INTERVENTIONS:
Diagnostic Test: Papanicolaou cytological test — Cervical smear stained using conventional Papanicolaou technique.
Diagnostic Test: Local cytological test (H&E stain) — Cervical smear stained using conventional hematoxylin and eosin staining techniques
Diagnostic Test: Validated HPV DNA Test — Digene HC2 HPV DNA Test
Diagnostic Test: Local HPV test — RealBest DNA HPV HR genotype (differential detection of human papillomavirus types 16, 18, 31, 33, 35, 39, 45, 51, 52, 56, 58, 59 DNA)
Diagnostic Test: Colposcopy — Women with positive cytology results are referred to colposcopy and biopsy
  Groups: High risk group

SUMMARY:
This single-institution cross-sectional non-inferiority validation study evaluates alternative techniques and tests for primary cervical cancer screening programs in Russia, particularly: local cytology staining techniques, local HPV tests.

DETAILED DESCRIPTION:
Cervical cytology practices are different across the world. While the Pap test became the cornerstone of the highly-effective cervical cancer screening in the countries that initially implemented population-based programs in the 60s and the 70s, alternative staining techniques were implemented in the Soviet Union. The tradition to apply other staining techniques than conventional Pap test remained unchanged in the national screening program implemented in the 2010s in Russia. As a new alternative option HPV testing showed effectiveness in screening women older than 30. The acceptable sensitivity and specificity of a screening test are crucial in population-based screening, that is why validation against "the gold standard" should be the first step in the process of program implementation. The objective of this study is to evaluate alternative techniques and tests for primary cervical cancer screening programs in Russia, particularly: local cytology staining techniques, local HPV tests in the population of 25-65 yo women without prior history of malignancy referred to colposcopy enriched with a population sample of women from several primary healthcare facilities referred to a primary screening test.

ELIGIBILITY:
Inclusion Criteria:

Age between 25 and 65 years old Referral to colposcopy or to a primary screening test Signed informed consent

Exclusion Criteria:

Prior history of malignancy or cervical dysplasia Prior history of cervical dysplasia

Ages: 25 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Gender identity
Study Population: 25-65 year-old women without prior history of malignancy referred to colposcopy enriched with a population sample of women from several primary healthcare facilities.
Sampling Method: Non-Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2020-07-13 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2023-07-01 (Estimated)

PRIMARY OUTCOMES:
Sensitivity | 24 months
  Cervical screening tests sensitivity
Specificity | 24 months
  Cervical screening tests specificity

SECONDARY OUTCOMES:
HPV prevalence by type | 24 months
  HPV prevalence by type based on genotyping in the population sample
Cervical dysplasia prevalence | 24 months
  Prevalence of cervical dysplasia in the population sample

OTHER OUTCOMES:
Safety of cervical smear | 24 months
  Adverse events after cervical smear
Safety of colposcopy and biopsy | 24 months
  Adverse events after colposcopy and biopsy

CONTACTS AND LOCATIONS:
Locations (1):
- N.N. Petrov National Medical Research Center of Oncology, Saint Petersburg, Russia

IPD SHARING:
Plan to Share IPD: Undecided